CLINICAL TRIAL: NCT03595865
Title: Efficacy of Tafluprost as an Adjunct to Medical Therapy for Residual Primary Open Angle Glaucoma and Residual Primary Angle-closure Glaucoma After Trabeculectomy
Brief Title: Efficacy of Tafluprost as an Adjunct to Medical Therapy for Residual Glaucoma After Trabeculectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: wangdabo (Other)
Responsible Party: Sponsor-Investigator, wangdabo, Principal Investigator, The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPLS2018G
Record Dates: First submitted 2018-05-25; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Glaucoma; Drugs
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- residual primary open angle glaucoma (Experimental): Each eye will be preformed tafluprostin 0.0015% at 9 PM, 1 time daily for 6months
  Interventions: Drug: tafluprostin
- residual primary angle-closure glaucoma (Experimental): Each eye will be preformed tafluprostin 0.0015% at 9 PM, 1 time daily for 6months
  Interventions: Drug: tafluprostin

INTERVENTIONS:
Drug: tafluprostin — Both patients in PACG and POAG groups will dose 1 time daily in each eye for 6months. Each eye will be preformed tafluprostin 0.0015% at 9 PM.

SUMMARY:
A 6-month, parallel-group study of the safety and efficacy of tafluprostin for Chinese patients with posttrabeculectomy residual primary angle-closure glaucoma or posttrabeculectomy residual primary open angle glaucoma.

DETAILED DESCRIPTION:
Enroll 60 eyes with posttrabeculectomy glaucoma (30 eyes with posttrabeculectomy residual primary angle-closure glaucoma. 30 eyes with posttrabeculectomy residual primary open angle glaucoma). Inclusive at 9 AM at eligibility visit and previously undergone trabeculectomy at least 30 days before screening visit. Qualified patients had a mean intraocular pressure (IOP) between 21 and 35mm Hg. All patients had documented residual PACG/POAG after trabeculectomy, with inadequate IOP control in at least one eye.The right eye was selected if both eyes showed about the same IOP. The previous IOP-lowering drugs were washed out before using tafluprost. Because all of the eyes had critical IOP levels, the design of this study was open-label, with emphasis on IOP change. Both patients in PACG and POAG groups will dose 1 time daily in each eye for 6 months. Each eye will be preformed tafluprost 0.0015% at 9 PM.The investigator monitored compliance via review of bottles at each follow-up visit, and at the last visit the old bottles will be returned and the investigator will keep them for storage. Efficacy and safety evaluations will be conducted at months 1, 2, 3, 4, 5, and 6 after the start of tafluprost treatment.The IOP will be measured at 1, 2, 3, 4, 5, and 6 month visit. All IOP measurements are to be performed at about the same time of day (at 9 AM at each visit). IOP was measured by Goldmann tonometer. The IOP value was the mean of 3 consecutive measurements.A visual field examination with automated perimetry(Octopus 101) using a threshold program was performed at the screening visit. If the visual field examination has been carried out within 12 weeks before the screening visit, no additional visual filed examination is required at the screening visit. A visual field examination and RNFL(retina nerve fiber layer) examination are to be performed at screening and the last visit respectively by the same technician with the same protocol. Topical examination by slit lamp is to be performed to evaluate the anterior segment. Ophthalmoscope examinations will be performed at screening and the last visit to examine the vitreous body, retina, and optic nervehead.The efficacy of tafluprost therapy is to be evaluated by comparing the baseline IOP and the IOP at various intervals after the start of treatment, by ANOVA test. The comparison of two groups was estimated by t test. The difference of the time point IOP between the 2 groups was analyzed by X2 test.

ELIGIBILITY:
Inclusion Criteria:

undergone trabeculectomy at least 30 days a mean intraocular pressure (IOP) between 21 and 35mmHg documented residual PACG/POAG after trabeculectomy visual acuity was more than 0.1

Exclusion Criteria:

women who were of childbearing potential (not postmenopausal or surgically sterile), pregnant, or nursing previous ocular mechanical trauma ocular infection or ocular inflammation any abnormality preventing reliable applanation tonometry of either eye cannot be safely discontinued from use of all ocular hypotensive medication(s) for a minimum period of 5 days to a maximum period of 4 weeks best-corrected visual acuity worse than 1.0 logMAR in study eye wore contact lenses refractive surgery or intraocular surgery within past 3 months severe or serious hypersensitivity to prostaglandins, prostaglandin analogs, or to any components of the study medications severe, unstable, or uncontrolled cardiovascular, hepatic, or renal disease less than 1 month stable dosing regimen of any medication used on a chronic basis that could affect IOP use of steroid or nonsteroid anti-inflammatory drug within 1 month therapy with another investigational agent within the past 30 days with other abnormal ocular condition or symptom preventing the patient from participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
IOP | 6 months
  The IOP will be measured at 1, 2, 3, 4, 5, and 6 month visit. All IOP measurements are to be performed at about the same time of day (at 9 AM at each visit). After topical anesthesia and conjunctiva sac stained byfluorescence, IOP was measured by Goldmann tonometer. The IOP value was the mean of 3 consecutive measurements.